CLINICAL TRIAL: NCT05031377
Title: The Effects of a Cardiovascular Health Education Program on Community-dwelling Older Adults at Risk of Atherosclerotic Cardiovascular Diseases: A Pilot Randomized Controlled Trial
Brief Title: Effects of Cardiovascular Health Education Program on Community-dwelling Older Adults at Risk of ASCVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ASCVD_OlderAudlts
Record Dates: First submitted 2021-08-19; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Diseases; Healthy Lifestyle; Health Education
Keywords: Older Adults; Physical Activity; Atherosclerotic Cardiovascular Disease; Lifestyle Modification; Health Education
MeSH Terms: conditions — Cardiovascular Diseases; Health Education; Motor Activity; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: Integrated Intervention (Experimental): Receive an integrated exercise and cardiovascular health education programme (HE programme)
  Interventions: Behavioral: HE programme
- Control (Sham Comparator): Receive usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: HE programme — Participants will receive a 12-week integrated exercise and cardiovascular health education programme (HE programme) which is constructed based on self-efficacy theory. A booster intervention in the form of SMS messaging will be given from Week 1 to Week 12.
  Arms: Experimental Arm: Integrated Intervention
Behavioral: Usual care — Participants will receive usual care which primarily includes an education talk on basic health issues. Governmental health education leaflets will be provided for reference.
  Arms: Control

SUMMARY:
Despite older adults being exposed to an increased risk of atherosclerotic cardiovascular disease (ASCVD), they are generally underrepresented in cardiovascular prevention programmes. The aim of this study is to assess the feasibility of implementing an integrated exercise and cardiovascular health education programme (HE programme) on older adults at risk of ASCVD.

DETAILED DESCRIPTION:
The study is a two-arm pilot randomized controlled trial. (1) The control group will receive a basic lifestyle modification talk and governmental education leaflets. (2) The experimental group will receive an integrated exercise and health education programme (HE programme) based on self-efficacy theory. Physical activity level, exercise self-efficacy and ASCVD risk profile including blood pressure, cardiac endurance, and anthropometric outcomes will be investigated via physiological assessments, medical history-taking or questionnaires at baseline, Week 6, and Week 12. Meanwhile, study feasibility will be primarily evaluated in terms of programme acceptability, intervention integrity, recruitment rate and retention rate throughout the process and at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adults ≧60 years old
* Having at least one ASCVD risk factor
* Pass the cardiovascular fitness evaluation
* Able to write and read Chinese, and communicate in Cantonese;
* Possess a mobile phone and able to make use of the phone in reading SMS

Exclusion Criteria:

* Visually impaired, hearing impaired, or suffer from cognitive, psychiatric, or muscular disorder
* Having a history of attending similar cardiovascular prevention program
* Having a previous history of coronary heart disease or stroke

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity level (total score) | At baseline, at Week 6, and at Week 12
  The physical activity level will be measured by the Chinese Version of Physical Activity Scale for the Elderly (PASE-C). The total score (from zero to 400 or above) is quantified based on frequency values and weights for these activities. The higher the score, the higher the level of physical activity.
Physical activity level (classification of physical activity level) | At baseline, at Week 6, and at Week 12
  The physical activity level will be measured by the Chinese version of International Physical Activity Questionnaire-short form (IPAQ-C-short form). Participants are classified into "inactive", "minimally active" or "health enhancing physical activity (HEPA) active" based on their physical activity levels.

SECONDARY OUTCOMES:
Exercise self-efficacy | At baseline, at Week 6, and at Week 12
  Exercise self-efficacy will be measured via the Chinese version of Self-Efficacy for Exercise (SEE-C). The total score ranges from 0 to 90. The higher the score, the greater the exercise self-efficacy.
ASCVD risk profiles (Blood pressure, weight, height, BMI & waist circumference, heart rate) | At baseline, at Week 6, and at Week 12
  The ASCVD risk profiles will be assessed by physical evaluations carried out by blinded, trained outcome assessors.
ASCVD risk profiles (2-minute walk test) | At screening stage, at Week 6, and at Week 12
  2-minute walk test will be adopted to examine aerobic capacity and self-paced walking capacity by measuring the walking distance covered at two minutes. It will be assessed by blinded, trained outcome assessors.
Acceptability of the program to participants | At Week 12
  It will be measured by a self-developed questionnaire
Acceptability of the program to outcome assessors | After the outcome assessors have finished their duties
  It will be measured by a self-developed questionnaire completed by outcome assessors
Acceptability of the program to lecture deliverers | After the lecture deliverers have finished their duties
  It will be measured by a self-developed questionnaire completed by lecture deliverers
Adverse events throughout the program | Throughout the study period
  Unfavorable or unintended events regarding the programme reported by participants throughout the study period.
Program safety evaluated by participants | At Week 12
  It will be measured via a self-developed questionnaire completed by participants
Eligibility rate | At baseline
  The number of eligible potential participants divided by the number of screened people
Recruitment rate | At baseline
  The percentage of participants who consent to join the study and being recruited
Retention rate | At baseline, at Week 6 and at Week 12
  The percentage of participants remaining in the study
Lecture attendance rate | Immediately after education session
  * The number of participants in the control group who attend the education talk divided by the number of participants who are randomized into the control group
  * The number of participants in the experimental group who attend the education session divided by the number of participants who are randomized into the experimental group
  * The number of participants in the two groups who attend the education session divided by the number of randomized participants
Adherence to intervention | At Week 6 and at Week 12
  * The number of participants in the experimental group who practice the tailor-made exercise learned during the intervention divided by the number of participants in the experimental group
  * Experimental group's frequency in performing tailor-made exercise related to the recommended exercise dosage
Attendance rate to data collection | At baseline, at Week 6 and at Week 12
  * The number of participants in the control group who attend the data collection divided by the number of participants who are randomized into the control group
  * The number of participants in the experimental group who attend the data collection divided by the number of participants who are randomized into the experimental group
  * The number of participants who attend the data collection divided by the number of randomized participants
Questionnaire completion rate | At baseline, at Week 6 and at Week 12
  The number of participants who complete the questionnaire divided by the number of distributed questionnaires
Missing data | At baseline, at Week 6 and at Week 12
  The percentage of missing data
Structured questionnaire | At baseline
  The questionnaire will primarily include patient demographics, medical history, lifestyle patterns, medication use and physical fitness evaluation data, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, PhD, Study Director — The Hong Kong Polytechnic University